CLINICAL TRIAL: NCT01236079
Title: Inpatient Technology-Supported Assisted Referral
Brief Title: Cessation Service Use and Effectiveness for Hospitalized Smokers
Acronym: I-TSAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Oregon Health and Science University (Other); Legacy Health System (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1U01HL105231-01 (NIH); 1U01HL105231-01 (NIH)
Record Dates: First submitted 2010-10-07; First posted 2010-11-08 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Assisted Referral & IVR (Experimental)
  Interventions: Behavioral: Assisted referral & IVR
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Assisted referral & IVR — includes assistance in enrolling in outpatient cessation services, pharmacy orders for cessation medication, interactive voice recognition follow-up
  Other Names: pharmacologic treatment, interactive voice recognition follow-up calls
  Arms: Assisted Referral & IVR

SUMMARY:
The goal of this patient-randomized effectiveness trial is to demonstrate that an inpatient technology-supported assisted referral (I-TSAR) and follow-up approach is an effective and cost-effective method to help hospitalized patients successfully quit smoking. The proposed study represents a unique opportunity to assess the effectiveness and cost-effectiveness of linking inpatient and outpatient delivery of smoking cessation services in two large and very different health care delivery systems. We will enroll 900 participants (600 intervention, 300 controls) over 15-months and collect follow-up survey and health care utilization data over 12 months to estimate: 1) smoking abstinence at 6 and 12 months for I-TSAR intervention recipients compared to usual care; 2) the dose effect on smoking abstinence at 6 and 12 months for I-TSAR recipients compared to usual care; 3) total and mean costs per participant for I-TSAR and usual care recipients, and, if effective, estimate the incremental cost-effectiveness of the intervention vs. controls at 12 months from health plan/insurer and societal perspectives; and 4) differences in health care utilization at 12 months for I-TSAR versus controls.

DETAILED DESCRIPTION:
The goal of this patient-randomized effectiveness trial is to demonstrate that an inpatient technology-supported assisted referral (I-TSAR) and follow-up approach is an effective and cost-effective method to help hospitalized patients successfully quit smoking. The proposed study represents a unique opportunity to assess the effectiveness and cost-effectiveness of linking inpatient and outpatient delivery of smoking cessation services in two large and very different health care delivery systems. We will enroll 900 participants (600 intervention, 300 controls) over 15-months and collect follow-up survey and health care utilization data over 12 months to estimate: 1) smoking abstinence at 6 and 12 months for I-TSAR intervention recipients compared to usual care; 2) the dose effect on smoking abstinence at 6 and 12 months for I-TSAR recipients compared to usual care; 3) total and mean costs per participant for I-TSAR and usual care recipients, and, if effective, estimate the incremental cost-effectiveness of the intervention vs. controls at 12 months from health plan/insurer and societal perspectives; and 4) differences in health care utilization at 12 months for I-TSAR versus controls.

This innovative study will provide important evidence for the effectiveness and cost effectiveness of technologically supporting hospital-based tobacco treatment specialists' efforts to provide treatment assistance to smokers interested in quitting and arrange for telephone follow-up support. The Tobacco Treatment Specialists will identify and enroll into the study smokers and recent quitters (ages 18 and over) admitted to KSMC and OHSU inpatient units, and randomize participants into usual care and I-TSAR intervention arms. Patients enrolled into the treatment arm will receive information about existing tobacco cessation programs and medications, will be enrolled into the cessation program and medication of their choice while admitted, and will be enrolled to receive four post-discharge follow-up calls over 7 weeks using an automated interactive voice recognition program developed with and provided by Eliza Corp. The Tobacco Treatment Specialist will work with hospital staff to initiate pharmacy orders for cessation medications, and coordinate cessation treatment with the participants' usual source of primary care (provider or clinic). Study staff will also work with hospital staff and managers to develop periodic clinic enrollment feedback reports.

Testing the approach in two different health care systems will provide generalized data for other health plans and insurers about the value of using electronic medical records systems to help inpatient staff facilitate smoking cessation treatment after discharge.

ELIGIBILITY:
Inclusion Criteria:

* willing to remain abstinent post discharge
* 1 cpd past 30 days
* active phone
* has a usual source of care
* willing to participate
* willing to provide contact information for follow up
* provide informed consent

Exclusion Criteria:

* critical care or labor/delivery units
* pregnant or breastfeeding
* physically unable to participate
* cognitively impaired
* no phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2011-12; Primary Completion 2013-11 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Fellows, PhD, Principal Investigator — Kaiser Permanente
Locations (3):
- United States (3):
  - Kaiser Permanente Sunnyside, Clackamas, Oregon
  - Legacy Emanuel Hospital, Portland, Oregon
  - Oregon Health & Science Univeristy, Portland, Oregon

REFERENCES:
- [Derived] Fellows JL, Mularski RA, Leo MC, Bentz CJ, Waiwaiole LA, Francisco MC, Funkhouser K, Stoney CM. Referring Hospitalized Smokers to Outpatient Quit Services: A Randomized Trial. Am J Prev Med. 2016 Oct;51(4):609-19. doi: 10.1016/j.amepre.2016.06.014. PMID 27647061
- [Derived] Duffy SA, Cummins SE, Fellows JL, Harrington KF, Kirby C, Rogers E, Scheuermann TS, Tindle HA, Waltje AH; Consortium of Hospitals Advancing Research on Tobacco (CHART). Fidelity monitoring across the seven studies in the Consortium of Hospitals Advancing Research on Tobacco (CHART). Tob Induc Dis. 2015 Sep 3;13(1):29. doi: 10.1186/s12971-015-0056-5. eCollection 2015. PMID 26336372
- [Derived] Fellows JL, Mularski R, Waiwaiole L, Funkhouser K, Mitchell J, Arnold K, Luke S. Health and economic effects from linking bedside and outpatient tobacco cessation services for hospitalized smokers in two large hospitals: study protocol for a randomized controlled trial. Trials. 2012 Aug 1;13:129. doi: 10.1186/1745-6215-13-129. PMID 22853325